CLINICAL TRIAL: NCT07242898
Title: Clinically Important or Just Statistically Significant? Minimal Clinically Important Difference for DVISS and PIN-Q in Children With Urinary Incontinence
Brief Title: Clinically Important or Just Statistically Significant? MCID for DVISS and PIN-Q in Children With UI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Artvin Coruh University (Other)
Responsible Party: Principal Investigator, Zeynep Yıldız Kızkın, Lecturer, Artvin Coruh University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCID-3
Record Dates: First submitted 2025-11-15; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Urinary Incontinence
Keywords: minimal clinically important difference; urinary incontinence; quality of life; ROC curve
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Intervention Model Description: In this prospective study, one treatment group was formed to receive SU.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Standard urotherapy (SU) (Experimental): Children with UI will receive SU as previously recommended.
  Interventions: Other: Standard Urotherapy (SU)

INTERVENTIONS:
Other: Standard Urotherapy (SU) — SU will be included appropriate provision of information and demystification, lifestyle advice, instructions, behavioral modifications to achieve optimal bladder and bowel habits, registration of symptoms and voiding habits, support, and encouragement

SUMMARY:
The goal of this study was to determine the Minimal Clinically Important Difference (MCID) for the Dysfunctional Voiding and Incontinence Symptom Score (DVISS) and the Pediatric Incontinence Questionnaire (PIN-Q) in children with urinary incontinence (UI).

DETAILED DESCRIPTION:
100 children with UI will receive standard urotherapy (SU) for 8 weeks. UI-related symptoms and quality of life (QoL) will be assessed with the DVISS and PIN-Q baseline and after treatment. The receiver operating characteristic (ROC) analysis and the Gamma coefficient will be employed to assess responsiveness.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of UI according to the International Children's Continence Society (ICCS) Guideline,
* children aged 5-13 years (when UI becomes more prevalent in children).

Exclusion Criteria:

* congenital anomalies of the uro-genital system,
* only neurogenic bladder dysfunction.

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2026-09-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Dysfunctional Voiding and Incontinence Symptom Score (DVISS) | Baseline
  DVISS includes 14 items: 13 assess lower urinary tract symptoms (LUTS), voiding and defecation habits day and night, and one evaluates impact on severity and daily life activities (DLA). A score of 8.5+ indicates abnormal voiding; higher scores mean more severe disease.
Dysfunctional Voiding and Incontinence Symptom Score (DVISS) | At Week 8, immediately after completion of the 8-week intervention
  DVISS includes 14 items: 13 assess lower urinary tract symptoms (LUTS), voiding and defecation habits day and night, and one evaluates impact on severity and daily life activities (DLA). A score of 8.5+ indicates abnormal voiding; higher scores mean more severe disease.

SECONDARY OUTCOMES:
Pediatric Urinary Incontinence Quality of Life Questionnaire (PIN-Q) | Baseline
  This 4-point Likert scale assesses the emotional impact of UI on a child, with 20 questions and a maximum score of 80. Higher scores mean a greater impact on QoL: 0-20 is mild, 21-50 moderate, and 51+ severe.
Pediatric Urinary Incontinence Quality of Life Questionnaire (PIN-Q) | At Week 8, immediately after completion of the 8-week intervention
  This 4-point Likert scale assesses the emotional impact of UI on a child, with 20 questions and a maximum score of 80. Higher scores mean a greater impact on QoL: 0-20 is mild, 21-50 moderate, and 51+ severe.

OTHER OUTCOMES:
Global Rating Change (GRC) | At Week 8, immediately after completion of the 8-week intervention
  The GRC comprised seven responses, ranging from 1 to 5, indicating "very much better," "slightly better," "no change," "slightly worse," and "very much worse," respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Yıldız Kızkın, Principal Investigator — Artvin Coruh University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Watanabe Y, Ikeda H, Ono T, Oyake C, Endo S, Onuki Y, Fuyama M, Watanabe T. Prevalence of Urinary Incontinence and Its Association With Neurodevelopmental Disorders Among Children in Japan. Neurourol Urodyn. 2025 Feb;44(2):458-463. doi: 10.1002/nau.25637. Epub 2024 Dec 9. PMID 39648965
- [Background] Shrestha N, Sahukhala S, K C D, Sandalcidi D, Adhikari SP. Prevalence of Urinary Incontinence in School Going Children: A Cross-sectional Study. J Nepal Health Res Counc. 2021 Jan 21;18(4):676-680. doi: 10.33314/jnhrc.v18i4.2506. PMID 33510509
- [Background] Linde JM, Nijman RJM, Trzpis M, Broens PMA. Prevalence of urinary incontinence and other lower urinary tract symptoms in children in the Netherlands. J Pediatr Urol. 2019 Apr;15(2):164.e1-164.e7. doi: 10.1016/j.jpurol.2018.10.027. Epub 2018 Nov 8. PMID 30583907
- [Background] Nieuwhof-Leppink AJ, Hussong J, Chase J, Larsson J, Renson C, Hoebeke P, Yang S, von Gontard A. Definitions, indications and practice of urotherapy in children and adolescents: - A standardization document of the International Children's Continence Society (ICCS). J Pediatr Urol. 2021 Apr;17(2):172-181. doi: 10.1016/j.jpurol.2020.11.006. Epub 2020 Nov 5. PMID 33478902
- [Background] Tekgul S, Stein R, Bogaert G, Undre S, Nijman RJM, Quaedackers J, 't Hoen L, Kocvara R, Silay MS, Radmayr C, Dogan HS. EAU-ESPU guidelines recommendations for daytime lower urinary tract conditions in children. Eur J Pediatr. 2020 Jul;179(7):1069-1077. doi: 10.1007/s00431-020-03681-w. PMID 32472266
- [Background] Malhotra NR, Kuhlthau KA, Rosoklija I, Migliozzi M, Nelson CP, Schaeffer AJ. Children's experience with daytime and nighttime urinary incontinence - A qualitative exploration. J Pediatr Urol. 2020 Oct;16(5):535.e1-535.e8. doi: 10.1016/j.jpurol.2020.10.002. Epub 2020 Oct 18. PMID 33148456
- [Background] Nacif A, de Abreu GE, Bessa Junior J, Veiga ML, Barroso U. Agreement between the visual analogue scale (VAS) and the dysfunctional voiding scoring system (DVSS) in the post-treatment evaluation of electrical nerve stimulation in children and adolescents with overactive bladder. J Pediatr Urol. 2022 Dec;18(6):740.e1-740.e8. doi: 10.1016/j.jpurol.2022.07.032. Epub 2022 Aug 3. PMID 36123285
- [Background] Thibodeau BA, Metcalfe P, Koop P, Moore K. Urinary incontinence and quality of life in children. J Pediatr Urol. 2013 Feb;9(1):78-83. doi: 10.1016/j.jpurol.2011.12.005. Epub 2012 Jan 10. PMID 22236468
- [Background] Husted JA, Cook RJ, Farewell VT, Gladman DD. Methods for assessing responsiveness: a critical review and recommendations. J Clin Epidemiol. 2000 May;53(5):459-68. doi: 10.1016/s0895-4356(99)00206-1. PMID 10812317
- [Background] Nieuwhof-Leppink AJ, Schroeder RPJ, van de Putte EM, de Jong TPVM, Schappin R. Daytime urinary incontinence in children and adolescents. Lancet Child Adolesc Health. 2019 Jul;3(7):492-501. doi: 10.1016/S2352-4642(19)30113-0. Epub 2019 May 4. PMID 31060913
- [Background] Akbal C, Genc Y, Burgu B, Ozden E, Tekgul S. Dysfunctional voiding and incontinence scoring system: quantitative evaluation of incontinence symptoms in pediatric population. J Urol. 2005 Mar;173(3):969-73. doi: 10.1097/01.ju.0000152183.91888.f6. PMID 15711352
- [Background] Frawley H, Shelly B, Morin M, Bernard S, Bo K, Digesu GA, Dickinson T, Goonewardene S, McClurg D, Rahnama'i MS, Schizas A, Slieker-Ten Hove M, Takahashi S, Voelkl Guevara J. An International Continence Society (ICS) report on the terminology for pelvic floor muscle assessment. Neurourol Urodyn. 2021 Jun;40(5):1217-1260. doi: 10.1002/nau.24658. Epub 2021 Apr 12. PMID 33844342
- [Background] Greco NJ, Anderson AF, Mann BJ, Cole BJ, Farr J, Nissen CW, Irrgang JJ. Responsiveness of the International Knee Documentation Committee Subjective Knee Form in comparison to the Western Ontario and McMaster Universities Osteoarthritis Index, modified Cincinnati Knee Rating System, and Short Form 36 in patients with focal articular cartilage defects. Am J Sports Med. 2010 May;38(5):891-902. doi: 10.1177/0363546509354163. Epub 2009 Dec 31. PMID 20044494
- [Background] Lehman LA, Velozo CA. Ability to detect change in patient function: responsiveness designs and methods of calculation. J Hand Ther. 2010 Oct-Dec;23(4):361-70; quiz 371. doi: 10.1016/j.jht.2010.05.003. Epub 2010 Jul 17. PMID 20638823